CLINICAL TRIAL: NCT00210899
Title: A Phase III, Randomized, Double-Blind Study of Ceftobiprole Versus Comparator in the Treatment of Complicated Skin and Skin Structure Infections
Brief Title: Ceftobiprole in the Treatment of Resistant Staphylococcus Aureus Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR005029; BAP00414 (Other: Basilea Pharmaceutica Ltd.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Skin Diseases, Infectious; Skin Diseases, Bacterial; Staphylococcal Skin Infections
Keywords: Complicated Skin Infections; Infectious Skin Diseases; Bacterial Skin Diseases; Staphylococcal Skin Infections; Cephalosporin
MeSH Terms: conditions — Skin Diseases, Infectious; Skin Diseases, Bacterial; Staphylococcal Skin Infections | interventions — ceftobiprole medocaril; Vancomycin; Ceftazidime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin plus Ceftazidime (Active Comparator): Vancomycin 1g q12h as 1h infusions plus Ceftazidime 1g q8h in 2h-infusions, 7-14d
  Interventions: Drug: Vancomycin plus Ceftazidime
- Ceftobiprole medocaril (Experimental): Ceftobiprole medocaril 500mg q8h as 2h infusions, 7-14d
  Interventions: Drug: ceftobiprole medocaril

INTERVENTIONS:
Drug: ceftobiprole medocaril
  Arms: Ceftobiprole medocaril
Drug: Vancomycin plus Ceftazidime
  Arms: Vancomycin plus Ceftazidime

SUMMARY:
The purpose of this study is to compare the clinical cure rate of ceftobiprole medocaril versus a comparator in the treatment of patients with complicated skin and skin structure infections. The study will also characterize the safety and tolerability of treatment with ceftobiprole medocaril in patients with complicated skin and skin structure infections.

DETAILED DESCRIPTION:
Ceftobiprole medocaril is a cephalosporin antibiotic with anti-MRSA (Methicillin-Resistant Staphylococcus Aureus) activity. Ceftobiprole medocaril is not yet approved for the treatment of complicated skin and skin structure infections. This is a randomized, double-blind, multicenter study of ceftobiprole medocaril plus placebo versus a comparator to assess the effectiveness and safety of ceftobiprole medocaril in patients with complicated skin and skin structure infections. The patients will be randomized to ceftobiprole medocaril plus placebo or a comparator. The patients can be treated as in-patient, out-patient, or through a home agency, at the discretion of the investigator. The primary endpoint is the clinical cure rate of ceftobiprole medocaril at the test-of-cure visit. The patients will receive either ceftobiprole medocaril plus placebo or a comparator for 7 to 14 days (unless extended at discretion of medical monitor).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an infection consistent with complicated skin and skin structure infections.

Exclusion Criteria:

* Known or suspected hypersensitivity to any study medication or other related anti-infective medication
* Any known or suspected condition or concurrent treatment contraindicated by the prescribing information
* Previous enrollment in this study
* Treatment with any investigational drug within 30 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate (the ratio of the number of clinically cured patients to the total number of patients in the population) at 7-14 days after the end of therapy. | 7 weeks
  7-14 days treatment, test of cure assessment at 7-14 days after end of treatment, late follow-up 28-35 days after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Noel GJ, Bush K, Bagchi P, Ianus J, Strauss RS. A randomized, double-blind trial comparing ceftobiprole medocaril with vancomycin plus ceftazidime for the treatment of patients with complicated skin and skin-structure infections. Clin Infect Dis. 2008 Mar 1;46(5):647-55. doi: 10.1086/526527. PMID 18225981
- See also: Ceftobiprole in the Treatment of Resistant Staphylococcus Aureus Skin and Skin Structure Infections — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=630&filename=CR005029_CSR.pdf